CLINICAL TRIAL: NCT03089138
Title: Efficacy and Safety of Regan Tangjiang for Treating the Common Cold With Wind-heat Syndrome: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo and Active-Controlled Phase 2b Study
Brief Title: Efficacy and Safety of Regan Tangjiang for Treating the Common Cold With Wind-heat Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Da-an Bio-technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: regan tangjiang phase 2
Record Dates: First submitted 2017-03-13; First posted 2017-03-24 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Cold
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regan Tangjiang，Simulation Shufengjiere Capsules (Experimental)
  Interventions: Drug: Regan Tangjiang
- Simulation Regan Tangjiang，Shufengjiere Capsules (Active Comparator)
  Interventions: Drug: Regan Tangjiang
- Simulation Regan Tangjiang and Shufengjiere Capsules (Placebo Comparator)
  Interventions: Drug: Regan Tangjiang

INTERVENTIONS:
Drug: Regan Tangjiang — The treatment duration is 3 consecutive days.

SUMMARY:
Efficacy and Safety of Regan Tangjiang for treating the common cold with wind-heat syndrome: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo and Active-Controlled Phase 2b Study

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of common cold according to Western Medicine，with symptoms onset and fever less than 24 hours prior to randomization；
* After the onset of the disease, with the following symptoms: sore throat and axillary temperature between 38.5 and 38.9°C inclusive.
* Diagnosis of wind-heat syndrome according to TCM；
* Aged between 18 to 65 years；
* Willingness to participate and to sign the informed consent form.

Exclusion Criteria:

* Participants with Pneumonia, suppurative tonsillitis, acute tracheobronchitis, acute and chronic sinusitis, pulmonary tuberculosis and other diseases;
* White blood cell count >11.0×109/L, or neutrophil percentage>75%;
* Participants with liver function 1.5 times higher than the normal upper limit or serum creatinine higher than the normal upper limit;
* Participants with severe primary diseases of cardiovascular, brain, lung, liver, kidney and hematopoietic system , such as viral hepatitis, hemophilia, diabetes, psychosis and so on;
* Participants who had used other drugs to treat common cold after the onset of the disease, including antivirals, antibiotics and traditional Chinese medicine.
* Women who are pregnant or breast-feeding;
* Allergic condition (refer to history of allergy to two or more drugs or food) or allergy to the drug composition(s);
* Participation in another clinical study of an investigational drug within 3 months
* Participants who are not suitable for the trial decided by the researchers for any reason, such as pregnancy, frequently changes in work or living environments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Time to fever relief | day 1 to day 3
  The median time from the first dosing to time when the body temperature drops by at least 0.5℃.In this study, all patients will be required to record their body temperature in the patient diary every 2 hours within the first 12 hours and every 4 hours during the following 12 hours. After that, it should be recorded four times at a fixed time every day.

SECONDARY OUTCOMES:
Time to fever clearance | day 1 to day 3
  The median time from the first dose administration to the time when the body temperature drops below 37.3℃ and lasts for 24 hours.
Time to symptom disappearance | day 1 to day 3
  The median time from study enrollment to the time when each individual symptom （such as fever, pharyngalgia, headache, runny nose, blocked nose, sneezing, cough） completely disappear.
Disappearance rate of symptoms | day 1 to day 3
  The percentage of patients with each individual symptom completely disappear from study enrollment to three days treatments.
Efficacy in TCM symptom and sign scores | day 1 to day 3
  The TCM symptom scoring system used in the study follows the Guidelines for Clinical Research of New Chinese Medicine, in which all symptoms are graded.
Usage of emergency medicines | day 1 to day 3
  Usage of emergency medicines is defined as the percentage of patients using emergency medicines (paracetamol).

IPD SHARING:
Plan to Share IPD: Undecided